CLINICAL TRIAL: NCT03289065
Title: Fabry Outcome Survey (FOS)
Acronym: FOS
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: FOS
Record Dates: First submitted 2017-08-17; First posted 2017-09-20 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Fabry Disease
Keywords: Genetic; Fabry Disease; Glycolipid; lysosomal
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FOS Participant: FOS is a disease registry open to all Fabry participants irrespective of treatment status or type of treatment.

SUMMARY:
The purpose of this study is to collect data that will increase understanding of Fabry disease history and progression, in treated and untreated patients with Fabry disease. The data from FOS may provide guidance to healthcare professionals about disease treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a documented diagnosis of Fabry disease

   * This may include a genetic mutation analysis. The collection of the genetic mutation analysis result is optional and dependent on the participant providing their consent for this data to be used in the FOS registry.
   * Participants can be untreated, currently or previously treated with Replagal, or any other approved treatment for Fabry disease.
2. Signed and dated written informed consent from the participant

   * For participants aged less than (<) 18 years (or as per local regulation), parent and/or participant's legally authorized representative (LAR), and assent of the minor, where applicable, is necessary.
   * If a participant is unable to read or if a legally acceptable representative is unable to read, an impartial witness should be present during the informed consent discussion and should sign and personally date the informed consent.
   * Informed consent must be obtained from LARs for cognitively impaired participants when applicable.

Exclusion Criteria:

1. Participants currently enrolled in ongoing blinded clinical trials (drugs or devices; includes all blinded trials) will be excluded from the Registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The FOS registry is open to participants with Fabry disease irrespective of their treatment. Participants may be untreated, currently treated or have been previously treated with Replagal, or any other approved treatment for Fabry disease. There is no predetermined sample size.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2001-04-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to year 20
  An adverse event (AE) is any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in the registry, whether or not considered product-related. This includes an exacerbation of a pre-existing condition. An AE or ADR that meets one or more of the following criteria/outcomes is classified as SAE whether considered to be related to the pharmaceutical product or not: death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalizations, a persistent or significant disability or incapacity, a congenital anomaly or birth defect and important medical events.
Number of Participants With Infusion-related Reactions (IRRs) | Baseline to year 20
  An infusion-related reaction (IRR) is defined as an AE that has been assessed as at least possibly related to treatment with Replagal and occurs during an infusion or up to 24 hours post Replagal infusion.
Renal Function by Estimated Glomerular Filtration Rate (eGFR) | Baseline to year 20
  Renal function will be measured by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) for adults and by Counahan-Barratt for children (<18 years).
Left Ventricular Mass Index (LVMI) | Baseline to year 20
  Left ventricular mass index (LVMI) will be assessed from baseline or from birth (age at event) to evaluate the course of Fabry disease in participants who are currently untreated or are being treated with an approved Fabry treatment.
Age at Mortality Event (survival) | Baseline to year 20
  Age at mortality event (survival) will be analysed with relevant split by demographic or baseline characteristic using Kaplan-Meier survival estimates with censoring at last visit in Fabry Outcome Survey (FOS)
Time to First Morbidity Event | Baseline to year 20
  Time to first morbidity event will be analysed with relevant split by demographic or baseline characteristic using Kaplan-Meier survival estimates with censoring at last visit in FOS.
Age at First Morbidity Event | Baseline to year 20
  Age at first morbidity event will be analysed with relevant split by demographic or baseline characteristic using Kaplan-Meier survival estimates with censoring at last visit in FOS.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Shire, Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Revel-Vilk S, Ramaswami U, Pintos-Morell G, Hughes D, Nicholls K, Reisin R, Giugliani R, Goker-Alpan O, Istaiti M, Gill A, Scarpa M, Botha J. Safety analysis of self-administered enzyme replacement therapy using data from the Fabry Outcome and Gaucher Outcome Surveys. Orphanet J Rare Dis. 2025 Mar 28;20(1):145. doi: 10.1186/s13023-024-03416-2. PMID 40155993
- [Derived] Beck M, Ramaswami U, Hernberg-Stahl E, Hughes DA, Kampmann C, Mehta AB, Nicholls K, Niu DM, Pintos-Morell G, Reisin R, West ML, Schenk J, Anagnostopoulou C, Botha J, Giugliani R. Twenty years of the Fabry Outcome Survey (FOS): insights, achievements, and lessons learned from a global patient registry. Orphanet J Rare Dis. 2022 Jun 20;17(1):238. doi: 10.1186/s13023-022-02392-9. PMID 35725623
- [Derived] Feriozzi S, Linhart A, Ramaswami U, Kalampoki V, Gurevich A, Hughes D; Fabry Outcome Survey Study Group. Effects of Baseline Left Ventricular Hypertrophy and Decreased Renal Function on Cardiovascular and Renal Outcomes in Patients with Fabry Disease Treated with Agalsidase Alfa: A Fabry Outcome Survey Study. Clin Ther. 2020 Dec;42(12):2321-2330.e0. doi: 10.1016/j.clinthera.2020.10.007. Epub 2020 Nov 17. PMID 33218740
- [Derived] Parini R, Pintos-Morell G, Hennermann JB, Hsu TR, Karabul N, Kalampoki V, Gurevich A, Ramaswami U; FOS Study Group. Analysis of Renal and Cardiac Outcomes in Male Participants in the Fabry Outcome Survey Starting Agalsidase Alfa Enzyme Replacement Therapy Before and After 18 Years of Age. Drug Des Devel Ther. 2020 Jun 3;14:2149-2158. doi: 10.2147/DDDT.S249433. eCollection 2020. PMID 32581513
- [Derived] Ramaswami U, Beck M, Hughes D, Kampmann C, Botha J, Pintos-Morell G, West ML, Niu DM, Nicholls K, Giugliani R; FOS Study Group. Cardio- Renal Outcomes With Long- Term Agalsidase Alfa Enzyme Replacement Therapy: A 10- Year Fabry Outcome Survey (FOS) Analysis. Drug Des Devel Ther. 2019 Oct 25;13:3705-3715. doi: 10.2147/DDDT.S207856. eCollection 2019. PMID 31749608